CLINICAL TRIAL: NCT00379795
Title: An Open-Label, Multicenter Extension Study to Evaluate the Safety and Tolerability of Ranibizumab in Subjects With Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (AMD) or Macular Edema Secondary to Retinal Vein Occlusion (RVO) Who Have Completed a Genentech-Sponsored Ranibizumab Study
Brief Title: An Extension Study to Evaluate the Safety and Tolerability of Ranibizumab in Subjects With Choroidal Neovascularization Secondary to AMD or Macular Edema Secondary to RVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF3426g (Cohort 1)
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Choroidal Neovascularization, Age-related Macular Degeneration
Keywords: CNV; Lucentis; AMD; Age-related macular degeneration; RVO
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Ranibizumab

ARMS (1):
- Ranibizumad 0.5 mg (Experimental): Ranibizumab 0.5 mg intravitreal injection 0.5 mg in the study eye on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment.
  Interventions: Drug: Ranibizumab 0.5 mg

INTERVENTIONS:
Drug: Ranibizumab 0.5 mg — Ranibizumab intravitreal injection 0.5 mg in a single-dose regimen given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year)

SUMMARY:
This was an open-label, multicenter, extension study of intravitreally administered ranibizumab in two cohorts. The first cohort (reported here) enrolled patients with primary or recurrent Choroidal Neovascularization (CNV) secondary to Age-Related Macular Degeneration (AMD) who completed the treatment phase of a Genentech sponsored study (FVF2598g (NCT00056836), FVF2587g (NCT00061594), or FVF2428g (NCT00056823)). The second cohort enrolled patients with macular edema secondary to Retinal Vein Occlusion (RVO) who completed the 6-month treatment and 6-month observation phases (12 months total) of a Genentech sponsored study (FVF4165g (NCT00486018) or FVF4166g (NCT00485836)). The results of the second cohort are reported separately (NCT01442064). The first cohort of this study enrolled two subsets of patients: ranibizumab experienced and ranibizumab-naive. Patients were enrolled within 14 days of completion of the 24 month treatment phase of the previous study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Completion of the treatment phase (through Month 24) of a Genentech-sponsored ranibizumab study for AMD (FVF2598g, FVF2587g, or FVF2428g) (Cohort 1)
* Expectation by the investigator that the subject may potentially benefit from intravitreal anti-vascular endothelial growth factor (VEGF) treatment

Exclusion Criteria:

* Previous subfoveal focal laser photocoagulation in the study eye
* Previous pegaptanib sodium injection in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1 month preceding Day 0 of this extension study
* History of submacular surgery or other surgical intervention for AMD in the study eye
* History of glaucoma filtering surgery in the study eye
* History of corneal transplant in the study eye
* Concurrent use of systemic anti-EGF agents
* Use of AMD treatments not approved by the FDA
* Use of intravitreal Avastin(R) (bevacizumab) in the study eye and/or fellow eye
* CNV in either eye due to other causes than AMD, such as ocular histoplasmosis, trauma, or pathologic myopia for Cohort 1
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 30 mmHg despite treatment with antiglaucoma medication)
* Pregnancy or lactation
* Premenopausal women not using adequate contraception
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications
* Current treatment for active systemic infection
* Inability to comply with study or follow-up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 853 (Actual)
Dates: Start 2005-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Tuomi, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open label multicenter extension study for participants who have completed one of the following studies: FVF2428g (NCT00056823), FVF2587g (NCT00061594) or FVF2598g (NCT0056823). Cohort 1 includes patients with Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (AMD).
Pre-assignment Details: Participants were classified according to ranibizumab exposure in the previous study and in the extension study. 63 participants (Untreated Group) did not receive study drug in this extension study or in the previous studies and are not included in the safety analyses.
Groups:
- RanibizumabTreated Initial Mono: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. Participants in this group received ranibizumab monotherapy (Mono) in previous studies, that is, ranibizumab alone in study FVF2598g or ranibizumab in combination with sham photodynamic therapy (PDT) in study FVF2587g.
- RanibizumabTreated Initial + PDT: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. This group includes participants who received ranibizumab in combination with photodynamic therapy in Study FVF2428g
- RanibizumabTreated Sham XO: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. Ranibizumab Treated Sham Crossover (XO) includes participants who received sham intravitreal injections before crossing over to receive ranibizumab intravitreal injections in study FVF2598g or this extension study.
- Ranibizumab Treated PDT XO: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. Ranibizumab Treated PDT XO includes participants who received sham intravitreal injections in combination with photodynamic therapy in study FVF2428g or study FVF2587g before crossing over to receive ranibizumab intravitreal injections in study FVF2428g, study FVF2587g or this study.
- Ranibizumab Untreated Group: In this extension study participants did not receive Ranibizumab. Participants in this group were enrolled in one of the following studies: FVF2428g (NCT00056823), FVF2587g (NCT00061594) FVF2598g (NCT0056823) but did not receive Ranibizumab intravitreal injections in that study or in this extension study (FVF3426g).
Period: Overall Study
Arm/Group | RanibizumabTreated Initial Mono | RanibizumabTreated Initial + PDT | RanibizumabTreated Sham XO | Ranibizumab Treated PDT XO | Ranibizumab Untreated Group
Started | 526 | 74 | 116 | 74 | 63
Received Ranibizumab in Extension Study | 377 | 41 | 113 | 55 | 0
Completed | 50 | 23 | 23 | 6 | 14
Not Completed | 476 | 51 | 93 | 68 | 49
Not completed — Death | 31 | 8 | 6 | 4 | 7
Not completed — Adverse Event | 17 | 3 | 3 | 1 | 4
Not completed — Lost to Follow-up | 8 | 1 | 2 | 1 | 4
Not completed — Physician Decision | 25 | 0 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 94 | 11 | 19 | 7 | 14
Not completed — Subject non-compliance | 7 | 2 | 0 | 0 | 1
Not completed — Verteporfin photodynamic therapy in eye | 3 | 0 | 0 | 1 | 0
Not completed — Subjects condition mandated intervention | 34 | 9 | 7 | 5 | 7
Not completed — Sponsor's decision | 257 | 17 | 54 | 47 | 10

BASELINE CHARACTERISTICS:
Groups:
- RanibizumabTreated Initial Mono: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. Participants in this group received ranibizumab 0.5 mg monotherapy, that is, ranibizumab alone in study FVF2598g or ranibizumab in combination with sham photodynamic therapy (PDT) in study FVF2587g.
- RanibizumabTreated Initial + PDT: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. This group includes participants who received ranibizumab 0.5 mg intravitreal injections in combination with photodynamic therapy in Study FVF2428g.
- RanibizumabTreated Sham XO: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. Ranibizumab Treated Sham Crossover (XO) includes participants who received sham intravitreal injections before crossing over to receive ranibizumab 0.5mg intravitreal injections in previous study FVF2598g or in this extension study.
- Ranibizumab Treated PDT XO: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. Ranibizumab Treated PDT XO includes participants who received sham intravitreal injections in combination with photodynamic therapy in study FVF2428g or study FVF2587g before crossing over to receive ranibizumab 0.5 mg intravitreal injections in previous studies FVF2428g, study FVF2587g or this extension study.
- Ranibizumab Untreated Group: In this extension study participants did not receive Ranibizumab. Participants in this group were previously enrolled in one of the following studies: FVF2428g (NCT00056823), FVF2587g (NCT00061594), FVF2598g (NCT0056823) but did not receive treatment with Ranibizumab in that study or in this extension study (FVF3426g).
- Total: Total of all reporting groups
Arm/Group | RanibizumabTreated Initial Mono | RanibizumabTreated Initial + PDT | RanibizumabTreated Sham XO | Ranibizumab Treated PDT XO | Ranibizumab Untreated Group | Total
Number analyzed (Participants) | 526 | 74 | 116 | 74 | 63 | 853
Age, Customized [Number; unit: participants]
  50 to < 65 | 29 | 5 | 5 | 8 | 4 | 51
  65 to < 75 | 117 | 19 | 27 | 21 | 10 | 194
  75 to < 85 | 277 | 42 | 61 | 35 | 29 | 444
  >= 85 | 103 | 8 | 23 | 10 | 20 | 164
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 42 | 76 | 41 | 36 | 499
  Male | 222 | 32 | 40 | 33 | 27 | 354

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ocular Adverse Events
Description: Number of participants with ocular adverse events in the following categories: any adverse events, serious adverse events, adverse events leading to study discontinuation, endophthalmitis and intraocular inflammation that occurred in the study eye (the eye that received all study drug injections) and the fellow eye (other eye).
  Only adverse events that occurred during this extension study are reported. For subjects in the crossover groups who started their first ranibizumab injection in this extension study, adverse events that occurred prior to any ranibizumab injection were also excluded.
Time Frame: 36 months
Population: All enrolled participants treated with Ranibizumab in this extension study or in one of the previous studies.
Measure: Number; unit: participants
Groups:
- Ranibizumab Treated Initial Mono: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. Participants in this group previously received ranibizumab monotherapy (Mono), that is, ranibizumab 0.5 mg intravitreal injection alone in previous study FVF2598g or ranibizumab 0.5 mg intravitreal injection in combination with sham photodynamic therapy (PDT) in previous study FVF2587g.
- Ranibizumab Treated Initial + PDT: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. This group includes participants who received ranibizumab 0.5 mg intravitreal injection in combination with photodynamic therapy in previous Study FVF2428g.
- Ranibizumab Treated Sham XO: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. Ranibizumab Treated Sham Crossover (XO) includes participants who received sham intravitreal injections before crossing over to receive ranibizumab 0.5 mg intravitreal injection in previous study FVF2598g or this extension study.
- Ranibizumab Treated PDT XO: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. Ranibizumab Treated PDT XO includes participants who received sham intravitreal injections in combination with photodynamic therapy in previous study FVF2428g or previous study FVF2587g before crossing over to receive ranibizumab 0.5 mg intravitreal injection in previous study FVF2428g, previous study FVF2587g or this extension study.
Arm/Group | Ranibizumab Treated Initial Mono | Ranibizumab Treated Initial + PDT | Ranibizumab Treated Sham XO | Ranibizumab Treated PDT XO
Number analyzed (Participants) | 526 | 74 | 116 | 74
participants
  Any adverse event in study eye | 418 | 56 | 96 | 59
  Serious adverse events in study eye | 46 | 2 | 6 | 2
  Adverse events led to discontinuation, study eye | 7 | 2 | 3 | 2
  Endophthalmitis in study eye | 1 | 0 | 0 | 0
  Intraocular inflammation in study eye, total | 8 | 2 | 4 | 1
  Serious Intraocular inflammation in study eye | 1 | 0 | 0 | 0
  Any adverse event in fellow eye | 304 | 50 | 72 | 47
  Serious adverse events in fellow eye | 22 | 4 | 6 | 3
  Adverse events led to discontinuation, fellow eye | 6 | 7 | 4 | 3
  Endophthalmitis in fellow eye | 0 | 0 | 0 | 0
  Intraocular inflammation in fellow eye, total | 5 | 0 | 0 | 0
  Serious intraocular inflammation in fellow eye | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Non-ocular Adverse Events
Description: Number of participants with non-ocular adverse events (not occurring in the eye) in the following categories: any adverse events, serious adverse events, adverse events leading to study discontinuation and death.
  Only adverse events that occurred during this extension study are reported. For subjects in the crossover groups who started their first ranibizumab injection in this extension study, adverse events that occurred prior to any ranibizumab injection were also excluded.
  Additional information about adverse events can be found in the adverse events section.
Time Frame: 36 months
Population: Enrolled participants treated with Ranibizumab in this extension study or in one of the previous studies.
Measure: Number; unit: participants
Arm/Group | Ranibizumab Treated Initial Mono | Ranibizumab Treated Initial + PDT | Ranibizumab Treated Sham XO | Ranibizumab Treated PDT XO
Number analyzed (Participants) | 526 | 74 | 116 | 74
participants
  Any non ocular adverse event | 427 | 61 | 92 | 58
  Serious non ocular adverse event | 169 | 21 | 33 | 20
  Non ocular adverse events led to discontinuation | 27 | 2 | 1 | 0
  Death | 31 | 8 | 6 | 4

3. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) at a Starting Test Distance of 2 Meters
Description: Change from baseline in Best corrected visual acuity (BCVA) was assessed by the number of letters a patient could read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) Eye Chart at a starting test distance of 2 meters. An increase in the number of letters read indicates improvement in visual acuity.
Time Frame: Extension study baseline, Months 3, 6, 9, 12, 15, 18, 21 and 24
Population: Enrolled participants. Observed data were used with no imputation. The number of participants for whom data was available for analyses is represented by "n".
Measure: Mean (Standard Deviation); unit: letters
Groups:
- Ranibizumab Initial Group: In this extension study participants received Ranibizumab injection 0.5 mg in a single-dose regimen given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Participants in this group were initially enrolled and received treatment with Ranibizumab in one of the following studies: FVF2428g (NCT00056823), FVF2587g (NCT00061594) or FVF2598g (NCT0056823).
- Ranibizumab Crossover Group: In this extension study participants received Ranibizumab injection 0.5 mg in a single-dose regimen given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Participants in this group were enrolled but did not initially receive Ranibizumab in Study FVF2428g (NCT00056823), Study FVF2587g (NCT00061594) or Study FVF2598g (NCT00056836) and then crossed over to receive Ranibizumab either in that initial study or this extension study.
- Ranibizumab Untreated Group: In this extension study participants did not receive Ranibizumab. Participants in this group were enrolled in one of the following studies: FVF2428g (NCT00056823), FVF2587g (NCT00061594) or FVF2598g (NCT0056823) but did not receive treatment with Ranibizumab in that study or this extension study.
- Total: All enrolled subjects
Arm/Group | Ranibizumab Initial Group | Ranibizumab Crossover Group | Ranibizumab Untreated Group | Total
Number analyzed (Participants) | 600 | 190 | 63 | 853
letters
  Change from Baseline at Month 3 (n=284, 84, 25) | -2.9 (8.9) | -2.9 (11.0) | 0.1 (6.6) | -2.7 (9.3)
  Change from Baseline at Month 6 (n=519, 149, 46) | -3.4 (8.8) | -1.6 (10.5) | 0.3 (7.0) | -2.8 (9.1)
  Change from Baseline at Month 9 (n=490, 149, 38) | -4.4 (10.8) | -1.7 (11.3) | -2.2 (7.5) | -3.7 (10.8)
  Change from Baseline at Month 12 (n=481, 142, 38) | -5.2 (11.1) | -2.3 (11.5) | -3.2 (8.0) | -4.5 (11.1)
  Change from Baseline at Month 15 (n=447, 138, 31) | -5.6 (10.8) | -2.2 (12.4) | -3.0 (8.9) | -4.7 (11.2)
  Change from Baseline at Month 18 (n=420, 135, 28) | -6.4 (11.9) | -2.0 (12.5) | -4.4 (9.5) | -5.3 (12.1)
  Change from Baseline at Month 21 (n=405, 129, 28) | -7.9 (13.0) | -2.1 (13.3) | -3.5 (10.8) | -6.3 (13.2)
  Change from Baseline at Month 24 (n=388, 127, 27) | -8.1 (13.0) | -2.0 (13.5) | -2.9 (8.5) | -6.4 (13.2)

4. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity at a Starting Test Distance of 4 Meters
Description: Change from baseline in Best corrected visual acuity (BCVA) was assessed by the number of letters a patient could read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) Eye Chart at a starting test distance of 4 meters. An increase in the number of letters read indicates improvement in visual acuity.
Time Frame: Extension study baseline, Months 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: letters
Groups:
- Ranibizumab Crossover Group: In this extension study participants received Ranibizumab injection 0.5 mg in a single-dose regimen given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Participants in this group were enrolled but did not initially receive Ranibizumab in Study FVF2428g (NCT00056823), Study FVF2587g (NCT00061594) or Study FVF2598g (NCT00056836) and then crossed over to receive Ranibizumab either in the initial study or this extension study.
Arm/Group | Ranibizumab Initial Group | Ranibizumab Crossover Group | Ranibizumab Untreated Group | Total
Number analyzed (Participants) | 600 | 190 | 63 | 853
letters
  Change from Baseline at Month 12 (n=446,133,35) | -5.4 (11.8) | -1.3 (11.8) | -3.2 (7.2) | -4.4 (11.7)
  Change from Baseline at Month 24 (n=352,122,25) | -7.5 (12.3) | -0.8 (13.0) | -3.1 (8.2) | -5.7 (12.7)

5. Primary Outcome: Number of Participants With Positive Serum Antibodies to Ranibizumab at Month 12 and Month 24
Description: Serum samples for the evaluation of antibodies to Ranibizumab were collected at Month 12 and Month 24 and were sent to a reference laboratory for analysis. If an injection of Ranibizumab was required at the visit, the samples were collected prior to the injection.
Time Frame: Month 12 and 24
Population: Population included all enrolled participants treated with Ranibizumab in the extension study or in one of the initial studies. The number of participants for whom data was available at Month 12 and Month 24 are represented by "n"
Measure: Number; unit: participants
Arm/Group | Ranibizumab Treated Initial Mono | Ranibizumab Treated Initial + PDT | Ranibizumab Treated Sham XO | Ranibizumab Treated PDT XO
Number analyzed (Participants) | 526 | 74 | 116 | 74
participants
  Month 12 (n=393,55,72,50) | 10 | 0 | 1 | 0
  Month 24 (n=316,45,78,42) | 9 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: The summary includes adverse events that occurred from enrollment in this extension study through 36 months (+/- 7 days).
Description: Safety Population includes all participants who received at least one dose of study drug in one of the initial studies or this extension study. As per the protocol participants who did not receive study drug were excluded from the analyses.
  Only adverse events that occurred during this extension study are reported.
Groups:
- Ranibizumab Treated Sham XO: In this extension study participants received Ranibizumab intravitreal injection 0.5 mg in the study eye given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Dosing interval was determined by the investigator, on the basis of clinical evaluations and judgment. Ranibizumab Treated Sham Crossover (XO) includes participants who received sham intravitreal injections before crossing over to receive ranibizumab 0.5 mg intravitreal injection in previous study FVF2428g or this extension study.
Arm/Group | Ranibizumab Treated Initial Mono | Ranibizumab Treated Initial + PDT | Ranibizumab Treated Sham XO | Ranibizumab Treated PDT XO
Serious Adverse Events (participants affected / at risk) | 213/526 | 26/74 | 43/116 | 24/74
Other Adverse Events (participants affected / at risk) | 491/526 | 70/74 | 110/116 | 71/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab Treated Initial Mono (N=526) | Ranibizumab Treated Initial + PDT (N=74) | Ranibizumab Treated Sham XO (N=116) | Ranibizumab Treated PDT XO (N=74)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 | 0 | 1 | 0
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 0
SICK SINUS SYNDROME (Cardiac disorders) | 1 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
HYPOPARATHYROIDISM (Endocrine disorders) | 1 | 0 | 0 | 0
MACULAR DEGENERATION (Eye disorders) | 21 | 2 | 5 | 1
CHOROIDAL NEOVASCULARISATION (Eye disorders) | 7 | 2 | 2 | 2
VISUAL ACUITY REDUCED (Eye disorders) | 11 | 1 | 0 | 0
RETINAL HAEMORRHAGE (Eye disorders) | 8 | 0 | 2 | 0
VITREOUS HAEMORRHAGE (Eye disorders) | 3 | 0 | 1 | 0
CATARACT (Eye disorders) | 3 | 0 | 0 | 0
MACULAR OEDEMA (Eye disorders) | 2 | 0 | 0 | 0
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 2 | 0 | 0 | 0
POSTERIOR CAPSULE OPACIFICATION (Eye disorders) | 1 | 0 | 1 | 0
RETINAL DEGENERATION (Eye disorders) | 2 | 0 | 0 | 0
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 1 | 0 | 0 | 0
PAPILLOEDEMA (Eye disorders) | 0 | 1 | 0 | 0
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 | 0 | 0 | 0
RETINAL PIGMENT EPITHELIAL TEAR (Eye disorders) | 1 | 0 | 0 | 0
SUBRETINAL FIBROSIS (Eye disorders) | 1 | 0 | 0 | 0
UVEITIS (Eye disorders) | 1 | 0 | 0 | 0
VITRITIS (Eye disorders) | 1 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 5 | 0 | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 0 | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0 | 0 | 0
ABDOMINAL COMPARTMENT SYNDROME (Gastrointestinal disorders) | 1 | 0 | 0 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 0 | 0 | 1
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
COLONIC STENOSIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DIVERTICULUM (Gastrointestinal disorders) | 1 | 0 | 0 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ILEUS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PHARYNGOESOPHAGEAL DIVERTICULUM (Gastrointestinal disorders) | 1 | 0 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CHEST PAIN (General disorders) | 4 | 0 | 1 | 1
DEATH (General disorders) | 2 | 0 | 1 | 0
ASTHENIA (General disorders) | 0 | 0 | 1 | 0
GRANULOMA (General disorders) | 1 | 0 | 0 | 0
HERNIA OBSTRUCTIVE (General disorders) | 1 | 0 | 0 | 0
IDIOSYNCRATIC DRUG REACTION (General disorders) | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 2 | 0 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 2 | 0 | 0 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 1 | 0 | 0 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 13 | 1 | 4 | 0
BRONCHITIS (Infections and infestations) | 5 | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 3 | 1 | 0 | 0
LOBAR PNEUMONIA (Infections and infestations) | 2 | 1 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 3 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 2 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 2 | 0 | 0 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0 | 1 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 1 | 0 | 0 | 0
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 | 0 | 0 | 0
KERATITIS HERPETIC (Infections and infestations) | 0 | 0 | 0 | 1
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1 | 0 | 0 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 0 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
UROSEPSIS (Infections and infestations) | 1 | 0 | 0 | 0
VIRAL MYOCARDITIS (Infections and infestations) | 1 | 0 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 8 | 1 | 1 | 1
FALL (Injury, poisoning and procedural complications) | 8 | 0 | 0 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
PUBIC RAMI FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
ARTERIAL INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
DEVICE FAILURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
MEDICATION ERROR (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
STRESS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
THERAPEUTIC AGENT TOXICITY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
INTRAOCULAR PRESSURE INCREASED (Investigations) | 2 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 | 0 | 1 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BLADDER CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OVARIAN EPITHELIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 6 | 1 | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 4 | 1 | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 3 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 2 | 0 | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 2 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 2 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 1 | 0 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 2 | 0 | 0 | 0
APHASIA (Nervous system disorders) | 1 | 0 | 0 | 0
BRAIN MASS (Nervous system disorders) | 1 | 0 | 0 | 0
BRAIN STEM INFARCTION (Nervous system disorders) | 0 | 1 | 0 | 0
CAROTID ARTERY DISEASE (Nervous system disorders) | 0 | 0 | 0 | 1
CEREBELLAR HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 1 | 0
CEREBRAL HAEMATOMA (Nervous system disorders) | 0 | 1 | 0 | 0
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 1 | 0 | 0 | 0
CONVULSION (Nervous system disorders) | 0 | 0 | 1 | 0
DEMENTIA (Nervous system disorders) | 1 | 0 | 0 | 0
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 | 0 | 0 | 0
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0 | 0 | 0
SPONDYLITIC MYELOPATHY (Nervous system disorders) | 1 | 0 | 0 | 0
THROMBOTIC STROKE (Nervous system disorders) | 1 | 0 | 0 | 0
BIPOLAR DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 2 | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 1 | 0 | 0 | 0
RENAL DISORDER (Renal and urinary disorders) | 1 | 0 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0 | 0
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 | 1 | 0 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
PELVIC PROLAPSE (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 1 | 3
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
AORTIC ANEURYSM (Vascular disorders) | 3 | 0 | 0 | 1
AORTIC STENOSIS (Vascular disorders) | 2 | 1 | 0 | 0
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 2 | 0 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 | 0 | 0 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0 | 1 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 1 | 0 | 1 | 0
ANEURYSM (Vascular disorders) | 1 | 0 | 0 | 0
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 1 | 0 | 0 | 0
AORTIC DISSECTION (Vascular disorders) | 1 | 0 | 0 | 0
HAEMORRHAGE (Vascular disorders) | 0 | 0 | 0 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 1 | 0 | 0 | 0
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 8 | 0 | 4 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 7 | 0 | 2 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 1 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 4 | 0 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 1 | 1 | 1
ANGINA PECTORIS (Cardiac disorders) | 2 | 1 | 0 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0 | 1 | 1
BRADYCARDIA (Cardiac disorders) | 1 | 1 | 0 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0 | 0 | 0
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab Treated Initial Mono (N=526) | Ranibizumab Treated Initial + PDT (N=74) | Ranibizumab Treated Sham XO (N=116) | Ranibizumab Treated PDT XO (N=74)
ANAEMIA (Blood and lymphatic system disorders) | 27 | 3 | 3 | 3
ATRIAL FIBRILLATION (Cardiac disorders) | 14 | 4 | 3 | 0
MACULAR DEGENERATION (Eye disorders) | 236 | 18 | 53 | 22
RETINAL HAEMORRHAGE (Eye disorders) | 197 | 21 | 47 | 31
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 124 | 20 | 33 | 17
CHOROIDAL NEOVASCULARISATION (Eye disorders) | 63 | 15 | 16 | 10
MACULAR OEDEMA (Eye disorders) | 70 | 6 | 15 | 8
CATARACT (Eye disorders) | 61 | 12 | 8 | 11
EYE PAIN (Eye disorders) | 56 | 4 | 13 | 8
MYODESOPSIA (Eye disorders) | 56 | 3 | 9 | 7
VISUAL ACUITY REDUCED (Eye disorders) | 32 | 4 | 3 | 4
DETACHMENT OF RETINAL PIGMENT EPITHELIUM (Eye disorders) | 33 | 3 | 12 | 3
MACULOPATHY (Eye disorders) | 30 | 4 | 4 | 5
VISION BLURRED (Eye disorders) | 31 | 4 | 5 | 2
EYE IRRITATION (Eye disorders) | 29 | 1 | 7 | 2
POSTERIOR CAPSULE OPACIFICATION (Eye disorders) | 29 | 1 | 6 | 2
FOREIGN BODY SENSATION IN EYES (Eye disorders) | 21 | 5 | 8 | 2
BLEPHARITIS (Eye disorders) | 25 | 5 | 3 | 2
EYE PRURITUS (Eye disorders) | 23 | 4 | 7 | 1
RETINAL DISORDER (Eye disorders) | 24 | 1 | 9 | 1
RETINAL DEGENERATION (Eye disorders) | 23 | 1 | 6 | 2
DRY EYE (Eye disorders) | 16 | 3 | 5 | 7
PHOTOPSIA (Eye disorders) | 14 | 4 | 3 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 31 | 5 | 5 | 9
NAUSEA (Gastrointestinal disorders) | 27 | 1 | 5 | 3
CONSTIPATION (Gastrointestinal disorders) | 22 | 0 | 6 | 1
NASOPHARYNGITIS (Infections and infestations) | 48 | 9 | 9 | 7
BRONCHITIS (Infections and infestations) | 43 | 3 | 7 | 4
URINARY TRACT INFECTION (Infections and infestations) | 38 | 3 | 8 | 3
INFLUENZA (Infections and infestations) | 25 | 2 | 5 | 4
SINUSITIS (Infections and infestations) | 22 | 4 | 7 | 2
EAR INFECTION (Infections and infestations) | 4 | 4 | 1 | 1
CONTUSION (Injury, poisoning and procedural complications) | 20 | 1 | 6 | 3
INTRAOCULAR PRESSURE INCREASED (Investigations) | 73 | 6 | 15 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 31 | 10 | 6 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 36 | 1 | 4 | 4
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 26 | 3 | 7 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 22 | 1 | 4 | 7
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 13 | 1 | 3 | 4
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 0 | 6 | 0
DEPRESSION (Psychiatric disorders) | 23 | 6 | 3 | 2
ANXIETY (Psychiatric disorders) | 23 | 5 | 2 | 2
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 7 | 2 | 2 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 15 | 1 | 2 | 4
HYPERTENSION (Vascular disorders) | 43 | 9 | 9 | 8
SUBMACULAR FLUID (Eye disorders) | 0 | 4 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No